CLINICAL TRIAL: NCT04370054
Title: Phase 3, Open-Label, Single-Arm Study to Evaluate the Efficacy and Safety of PF-07055480 (Recombinant AAV2/6 Human Factor VIII Gene Therapy) in Adult Male Participants With Moderately Severe to Severe Hemophilia A(FVIII:C≤1%)
Brief Title: Study to Evaluate the Efficacy and Safety of PF-07055480 / Giroctocogene Fitelparvovec Gene Therapy in Moderately Severe to Severe Hemophilia A Adults
Acronym: AFFINE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C3731003; 2024-512075-12-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2020-04-21; First posted 2020-04-30 (Actual); Results first posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-07

CONDITIONS: Hemophilia A
Keywords: PF-07055480; SB-525; Hemophilia; Factor VIII; FVIII; Gene Therapy; AAV; AAV6; Annualized bleeding rate; ABR; giroctocogene fitelparvovec; AFFINE
MeSH Terms: conditions — Hemophilia A | interventions — Genetic Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PF-07055480 (giroctocogene fitelparvovec) (Experimental): Single administration of PF-07055480
  Interventions: Biological: PF-07055480 (giroctocogene fitelparovec): Recombinant AAV2/6 Human Factor VIII Gene Therapy

INTERVENTIONS:
Biological: PF-07055480 (giroctocogene fitelparovec): Recombinant AAV2/6 Human Factor VIII Gene Therapy — Single IV infusion
  Other Names: Gene Therapy

SUMMARY:
C3731003 is a pivotal Phase 3 study to evaluate the clinical efficacy and safety of a single IV infusion of PF-07055480 / giroctocogene fitelparvovec (Recombinant AAV2/6 Human Factor VIII Gene Therapy) in adult male participants with moderately severe or severe hemophilia A (FVIII:C≤1%) for the study duration of 5 years. The study will enroll eligible participants who have been followed on routine prophylaxis with FVIII products in the Lead-In study C0371004.

ELIGIBILITY:
Main inclusion Criteria

* Males who have been followed on routine Factor VIII prophylaxis therapy during the lead-in study (C0371004) and have > = 150 documented exposure days to a Factor VIII protein product
* Moderately severe to severe hemophilia A (Factor VIII activity < =1%)
* Suspension of FVIII prophylaxis therapy post study drug infusion

Main exclusion Criteria

* Anti-AAV6 neutralizing antibodies
* History of inhibitor to Factor VIII
* Laboratory values at screening visit that are abnormal or outside acceptable study limits
* Significant and/or unstable liver disease, biliary disease, significant liver fibrosis
* Conditions associated with increased thromboembolic risk such as inherited or acquired thrombophilia, or a history of thrombotic events
* Planned surgical procedure requiring Factor VIII surgical prophylactic factor treatment 12 months from screening visit
* Active hepatitis B or C
* Serological evidence of human immunodeficiency virus HIV-1 or HIV-2 with Cluster of Differentiation 4 positive (CD4+) cell count ≤200 mm3 and/or viral load >20 copies/mL

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 77 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2028-10-25 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (36):
- United States (11):
  - NOW Physical Therapy, Mountain View, California
  - Clinical and Translational Research Unit (CTRU), Palo Alto, California
  - Lucile Packard Childrens Hospital, Palo Alto, California
  - Imaging Clinic at Stanford Medicine Outpatient Center in Redwood City, Redwood City, California
  - UCSF IDS Pharmacy, San Francisco, California
  - University of California, San Francisco - Clinical Research Center, San Francisco, California
  - University of California, San Francisco - Moffitt/Long Inpatient Hematology, San Francisco, California
  - University of California, San Francisco - Outpatient Hematology Clinic, San Francisco, California
  - Stanford Health Care, Stanford, California
  - Washington Institute for Coagulation, Seattle, Washington
  - University of Washington Medical Center - Translational Research Unit (TRU), Seattle, Washington
- The Alfred Hospital, Melbourne, Victoria, Australia
- Centro de Hematologia e Hemoterapia de Campinas - Hemocentro UNICAMP, Campinas, São Paulo, Brazil
- Canada (2):
  - McMaster University Medical Centre - Hamilton Health Sciences, Hamilton, Ontario
  - Juravinski Hospital - Hamilton Health Sciences, Hamilton, Ontario
- Hopital Necker, Paris, France
- Germany (2):
  - Vivantes Klinikum im Friedrichshain, Berlin
  - Klinikum der Johann Wolfgang Goethe-Universitaet, Medizinische Klinik II, Frankfurt am Main
- Greece (2):
  - General Hospital of Athens ''Laiko'', Athens, Attikí
  - General Hospital of Athens "Hippokration", Athens
- Italy (3):
  - Università degli studi di Roma "La Sapienza"- Policlinico Umberto I, Roma, RM
  - Azienda Ospedaliero Universitaria Careggi SODc Malattie Emorragiche e della Coagulazione, Florence
  - Dip. di Medicina Clinica e Chirurgia, Università degli Studi di Napoli Federico II - UOC di Medicina, Napoli
- Japan (2):
  - Nagoya University Hospital - Transfusion Medicine, Nagoya, Aichi-ken
  - Saitama Medical University Hospital, Iruma-gun, Saitama
- King Faisal Specialist Hospital & Research Center, Riyadh, Saudi Arabia
- Kyung Hee University Hospital at Gangdong, Seoul, South Korea
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - H.U. Rio Hortega, Valladolid
- Skåne University Hospital, Malmo, Skåne County, Sweden
- National Taiwan University Hospital, Taipei, Taiwan
- Turkey (Türkiye) (4):
  - Adana Acibadem Hospital, Adana
  - Gaziantep University Sahinbey Research and Training Hospital, Gaziantep
  - Ege University Medical Faculty, Pediatric Hematology, Izmir
  - Ege University Medical Faculty, Izmir
- Guy's and St. Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3731003

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with moderately severe to severe hemophilia A, who completed routine Factor VIII (FVIII) prophylaxis follow-up during the lead-in study C0371004 (NCT03587116), were enrolled in this study. Participants in this study received single infusion of PF-07055480/giroctocogene fitelparovec.
Pre-assignment Details: Results are presented for primary outcome measures and only those secondary outcome measures whose analysis was complete on a data cutoff date of 17 June 2024 (primary completion date [PCD]). Remaining outcome measures would be reported upon completion of their analyses at study completion date.
Groups:
- PF-07055480: Participants received a single infusion of PF-07055480 3.0*10^13 vector genomes per kilogram (vg/kg) intravenously on Day 1.
Period: Treatment Phase
Arm/Group | PF-07055480
Started | 77
Treated | 75
Completed | 75
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1
Period: Follow-Up Phase
Arm/Group | PF-07055480
Started | 75
Completed | 0
Not Completed | 75
Not completed — Ongoing | 75

BASELINE CHARACTERISTICS:
Population: The safety set included all participants enrolled in the study and who received the study intervention.
Groups:
- PF-07055480: Participants received a single infusion of PF-07055480 3.0*10^13 vg/kg IV on Day 1.
Arm/Group | PF-07055480
Number analyzed (Participants) | 75
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.27 (10.441)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 59
  Unknown or Not Reported | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 14
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 56
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Total Annualized Bleeding Rate (ABR)
Description: Bleeds for evaluation included both treated and untreated bleeds. Treated bleed: bleeding event necessitated administration of coagulation factor within 72 hours of signs or symptoms of bleeding. Untreated bleed: bleeding event did not necessitate administration of coagulation factor within 72 hours of signs and symptoms of bleeding. In this outcome measure total ABR following infusion of PF-07055480 in current study (post-infusion) and on prior FVIII prophylaxis regimen prior to infusion of PF-07055480 (pre-infusion, data collected from lead-in study C0371004) were reported. Total ABR for FVIII prophylaxis= [(Number of total bleeding episodes during pre-infusion period)*365.25]/ [(Number of days of follow-up in pre-infusion period)]. Total ABR for PF-07055480: [(Number of total bleeding episodes during post-infusion period)*365.25] / [(last date of post-infusion period - date of PF-07055480 infusion) - 77 days + 1].
Time Frame: FVIII Prophylaxis arm: a minimum of 7.4 months, up to maximum of 32.3 months (Pre-infusion period); PF-07055480 arm: Week 12 through at least 15 months of follow-up, maximum follow up was of 44.4 months (Post-infusion period)
Population: Efficacy analysis population included all participants in the 'Dosed' population [enrolled and received the study intervention] who completed at least 6 months of follow up in the lead-in study and at least 15 months of follow-up or discontinued from the study C3731003 prior to the data cutoff for reporting. Data within the same participants were compared between Pre and Post infusion (2 groups described below), with different specified periods/durations.
Measure: Mean (95% Confidence Interval); unit: Total bleeds per year
Groups:
- FVIII Prophylaxis: Participants who received FVIII prophylaxis replacement therapy during the lead-in study C0371004 and were enrolled to receive PF-07055480 infusion in current study C3731003. In this arm, data from participants for pre-infusion (of PF-07055480) from the lead-in study C0371004 period was included.
Arm/Group | FVIII Prophylaxis | PF-07055480
Number analyzed (Participants) | 50 | 50
Total bleeds per year | 4.73 [2.86 to 6.60] | 1.24 [-0.66 to 3.14]
Statistical Analysis 1: Comparison: FVIII Prophylaxis vs PF-07055480; A repeated measures GLM was used with bleeds as dependent variable in negative binomial distribution, an interaction of duration by treatment, and 'participant' as random and treatment & duration of follow-up as fixed effect; Test type: Non-Inferiority — A repeated measures negative binomial regression model was used to test non-inferiority with non-inferiority margin = 3 bleeds/year at the one-sided alpha level = 0.025; p = 0.0040, Generalized linear model (GLM) — One-sided p-value is reported; Mean Difference (Final Values) = -3.49, 95% CI 2-sided [-6.06 to -0.91] — Difference in mean = Mean PF-07055480 Total ABR - Mean FVIII Prophylaxis Total ABR

2. Secondary Outcome: Percentage of Participants With Coagulation FVIII Activity Levels Greater Than (>)5 Percent (%) at 15 Months
Description: FVIII activity level based on central laboratory chromogenic assay at Month 15
Time Frame: At 15 months following infusion of PF-07055480
Population: Efficacy analysis population included all participants in the 'Dosed' population [enrolled and received the study intervention] who completed at least 6 months of follow up in the lead-in study and at least 15 months of follow-up or discontinued from the study C3731003 prior to the data cutoff for reporting.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PF-07055480
Number analyzed (Participants) | 50
Percentage of participants | 84.00 [70.89 to 92.83]
Statistical Analysis 1: Comparison: PF-07055480; Test type: Superiority; p = 0.0086, One-sided exact binomial proportion test — One-sided p-value is reported

3. Secondary Outcome: Treated ABR
Description: Treated bleed was defined as an event which necessitated administration of coagulation factor within 72 hours of signs or symptoms of bleeding. In this outcome measure treated ABR following infusion of PF-07055480 in current study (post-infusion) and on prior FVIII prophylaxis regimen prior to infusion of PF-07055480 (pre-infusion, data collected from lead-in study C0371004) were reported. Treated ABR for FVIII prophylaxis= [(Number of treated bleeding episodes during pre-infusion period)*365.25]/ [(Number of days of follow-up in pre-infusion period)]. Treated ABR for PF-07055480: [(Number of treated bleeding episodes during post-infusion period)*365.25] / [(last date of post-infusion period - date of PF-07055480 infusion) - 77 days + 1].
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Treated bleeds per year
Arm/Group | FVIII Prophylaxis | PF-07055480
Number analyzed (Participants) | 50 | 50
Treated bleeds per year | 4.08 [2.52 to 5.64] | 0.07 [0.01 to 0.13]
Statistical Analysis 1: Comparison: FVIII Prophylaxis vs PF-07055480; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Repeated measures GLM — One-sided p-value is reported; Mean Difference (Final Values) = -4.01, 95% CI 2-sided [-5.57 to -2.45] — Difference in mean = Mean PF-07055480 Total ABR - Mean FVIII Prophylaxis Total ABR

4. Secondary Outcome: Annualized Infusion Rate (AIR) of Exogenous FVIII Activity
Description: AIR: [(Number of exogenous FVIII product infusions for any purpose during the given time period) * 365.25]/ (Number of days of follow-up in the given time period). In this outcome measure AIR of exogenous FVIII activity in current study (post-infusion) and on prior FVIII prophylaxis regimen prior to infusion of PF-07055480 (pre-infusion, data collected from lead-in study C0371004) were reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Exogenous infusions per year
Arm/Group | FVIII Prophylaxis | PF-07055480
Number analyzed (Participants) | 50 | 50
Exogenous infusions per year | 124.39 (53.882) | 0.21 (0.601)
Statistical Analysis 1: Comparison: FVIII Prophylaxis vs PF-07055480; Test type: Superiority; p < 0.0001, Paired t-test — One-sided p-value is reported; Mean Difference (Final Values) = -124.18, 95% CI 2-sided [-139.47 to 108.89] — Treatment Difference = (PF-07055480 AIR - FVIII Prophylaxis AIR)

5. Secondary Outcome: FVIII Activity Levels From Week 12 Through 15 Months Following PF-07055480 Infusion
Description: FVIII activity levels were assessed using chromogenic assay and one-stage clotting assay analyzed in the central laboratory. As pre-specified, for each participant, a geometric mean laboratory reading for FVIII activity was used to derived one single FVIII level by including all assessments from Week 12 through 15 months following PF-07055480 infusion; then mean and standard deviation as summary statistics was calculated across all evaluable participants and reported as data for this outcome measure. This resulting Factor VIII activity is expressed as percent of normal (%); which is used interchangeable with international unit per deciliter (IU/dL). "Normal Range" is typically considered 50-150% (or 50-150 IU/dL).
Time Frame: Week 12 through Month 15 following PF-07055480 Infusion
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of Normal
Arm/Group | PF-07055480
Number analyzed (Participants) | 50
Percentage of Normal
  Chromogenic Assay | 96.84 (90.521)
  One-Stage Assay | 134.95 (116.161)

6. Secondary Outcome: Annualized FVIII Consumption
Description: Annualized FVIII consumption was reported in international units per kilogram (IU/kg) and total units (in IU). This outcome measure compared data collected from lead-in study C0371004 and from current study C3731003. Data is reported in this outcome measure as mean of annualized FVIII consumption from all participants in this analysis population.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/kg
Arm/Group | FVIII Prophylaxis | PF-07055480
Number analyzed (Participants) | 50 | 50
IU/kg | 4082.7 (2291.90) | 6.6 (21.41)
Statistical Analysis 1: Comparison: FVIII Prophylaxis vs PF-07055480; Test type: Superiority; p < 0.0001, Paired t-test — One-sided p-value is reported; Mean Difference (Final Values) = -4076.06, 95% CI 2-sided [-4728.3 to -3423.8] — Treatment Difference (FVIII Consumption post-IP Infusion - FVIII Consumption during FVIII Prophylaxis)

7. Secondary Outcome: Total (Treated and Untreated) ABR Based on Cause
Description: Bleeds based on cause:spontaneous(bleeding for no apparent/known reason particularly into the joint,muscles and soft tissue)and traumatic(bleeding event occurring for an apparent/known reason).Bleeds related to a procedure/surgery such as hematomas/bruising which resulted from any surgeries or invasive procedure,or invasive diagnostic procedures were not counted as bleeds.Treated:necessitated administration of coagulation factor within 72hrs of sign or symptom of bleeding. Untreated:did not necessitate administration of coagulation factor within 72hrs of sign and symptom of bleeding.ABR for FVIII prophylaxis=[(Number of total bleeding episodes during pre-infusion)*365.25]/(Number of days of follow-up in pre-infusion period).ABR for PF-07055480[(Number of total bleeding episodes during post-infusion period)*365.25]/[(last date of post-infusion period-date of PF-07055480 infusion)-77 days+1].This outcome measure compared data collected from lead-inC0371004and from current studyC3731003.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Bleeds per year
Arm/Group | FVIII Prophylaxis | PF-07055480
Number analyzed (Participants) | 50 | 50
Bleeds per year
  Spontaneous | 3.27 (5.591) | 1.07 (6.540)
  Traumatic | 1.46 (3.416) | 0.14 (0.320)

8. Secondary Outcome: Treated ABR Based on Cause
Description: Bleeds based on cause were spontaneous (bleeding for no apparent/known reason particularly into the joint, muscles and soft tissues) and traumatic (bleeding event occurring for an apparent/known reason). Bleeds related to a procedure/surgery such as hematomas/bruising which resulted from any surgeries or invasive procedures, or invasive diagnostic procedure were not counted as bleeds. Treated: necessitated administration of coagulation factor within 72 hours of signs or symptoms of bleeding. Treated ABR for FVIII prophylaxis= [(Number of treated bleeding episodes during pre-infusion period)*365.25]/ (Number of days of follow-up in pre-infusion period). Treated ABR for PF-07055480: [(Number of treated bleeding episodes during post-infusion period)*365.25] /[(last date of post-infusion period - date of PF-07055480 infusion) - 77 days + 1]. This outcome measure compared data collected from lead-in study C0371004 and from current study C3731003.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Bleeds per year
Arm/Group | FVIII Prophylaxis | PF-07055480
Number analyzed (Participants) | 50 | 50
Bleeds per year
  Spontaneous | 2.81 (4.469) | 0.02 (0.119)
  Traumatic | 1.27 (3.270) | 0.07 (0.213)

9. Secondary Outcome: Total (Treated and Untreated) ABR Based on Location
Description: Target joint:major joint(hip,elbow,wrist,shoulder,knee&ankle)with repeated bleed(3 or more spontaneous bleed into a single joint within6month).Joint bleed:bleeding episode by rapid loss of motion as compared with baseline,associated with pain or unusual sensation,swelling&warmth over the joint.Muscle:bleeding episode into a muscle,determined by imaging study,associated with pain&or swelling &functional impairment.Treated:necessitated administration of coagulation factor within72hrs of sign or symptom of bleeding.Untreated:did not necessitate administration of coagulation factor within72hrs of sign&symptom of bleeding.FVIII prophylaxis=[(Number of total bleeding episodes during pre-infusion)*365.25]/(Number of days of follow-up in pre-infusion).PF-07055480:[(Number of total bleeding episodes during post-infusion)*365.25]/[(last date of post infusion-date of PF-07055480 infusion)-77days+1].This outcome measure compared data collected from lead-inC0371004 and from current studyC3731003.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Bleeds per year
Arm/Group | FVIII Prophylaxis | PF-07055480
Number analyzed (Participants) | 50 | 50
Bleeds per year
  All Joints | 3.28 (5.358) | 0.51 (2.819)
  Target Joints | 1.13 (4.026) | 0.02 (0.130)
  Soft Tissue/Muscle/Other | 1.55 (3.346) | 0.76 (4.303)

10. Secondary Outcome: Treated ABR Based on Location
Description: Target joint:major joint(hip,elbow,wrist,shoulder,knee,and ankle)with repeated bleeds(3 or more spontaneous bleeds into a single joint within 6month).Joint bleed:bleeding episode characterized by rapid loss of range of motion as compared with baseline,associated with pain or an unusual sensation in the joint,palpable swelling,and warmth of the skin over the joint.Muscle:bleeding episode into a muscle,determined clinically and/or by imaging study,associated with pain and/or swelling and functional impairment.Treated:necessitated administration of coagulation factor within72 hrs of sign or symptom of bleeding.FVIII prophylaxis=[(Number of treated bleeding episodes during pre-infusion)*365.25]/(Number of days of follow-up in pre-infusion).PF-07055480:[(Number of treated bleeding episodes during post-infusion)*365.25]/[(last date of post-infusion-date of PF-07055480 infusion)-77days+1].This outcome measure compared data collected from lead-in studyC0371004 and from current studyC3731003.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Bleeds per year
Arm/Group | FVIII Prophylaxis | PF-07055480
Number analyzed (Participants) | 50 | 50
Bleeds per year
  All Joints | 2.81 (4.449) | 0.06 (0.205)
  Target Joints | 0.88 (2.905) | 0.00 (0.000)
  Soft Tissue/Muscle/Other | 1.34 (2.985) | 0.03 (0.136)

11. Secondary Outcome: Percentage of Participants Without Bleeds
Description: Bleeds for evaluation included both treated and untreated bleeds. Treated bleed: necessitated administration of coagulation factor within 72 hours of signs or symptoms of bleeding. Untreated bleed: did not necessitate administration of coagulation factor within 72 hours of signs and symptoms of bleeding. In this outcome measure percentage of participants without bleeds following infusion of PF-07055480 in current study (post-infusion) and on prior FVIII prophylaxis regimen prior to infusion of PF-07055480 (pre-infusion) were reported. This outcome measure compared data collected from lead-in study C0371004 and from current study C3731003.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | FVIII Prophylaxis | PF-07055480
Number analyzed (Participants) | 50 | 50
Percentage of participants
  Without treated bleeds | 30 | 88
  Without treated and untreated bleeds | 26 | 64

12. Secondary Outcome: FVIII Activity Level at Weeks 24, 52, 65, and 104
Description: FVIII activity levels were assessed using chromogenic and one-stage clotting assay and which were analyzed in the central laboratory.
Time Frame: At Weeks 24, 52, 65 and 104
Population: Dosed analysis population included all participants enrolled in the study and who received the study intervention. Here "Number Analyzed" at each row represents the number of participants with valid FVIII assessments at the respective time points.
Measure: Mean (95% Confidence Interval); unit: Percentage of Normal
Arm/Group | PF-07055480
Number analyzed (Participants) | 75
Percentage of Normal
  Week 24: Chromogenic Assay | 101.59 [78.68 to 124.51]
  Week 24: One-Stage Assay | 147.14 [116.91 to 177.37]
  Week 52: Chromogenic Assay: number analyzed (Participants) | 55
  Week 52: Chromogenic Assay | 51.68 [37.67 to 65.69]
  Week 52: One-Stage Assay: number analyzed (Participants) | 55
  Week 52: One-Stage Assay | 80.14 [60.53 to 99.76]
  Week 65: Chromogenic Assay: number analyzed (Participants) | 49
  Week 65: Chromogenic Assay | 51.08 [35.51 to 66.65]
  Week 65: One-Stage Assay: number analyzed (Participants) | 49
  Week 65: One-Stage Assay | 73.99 [54.34 to 93.65]
  Week 104: Chromogenic Assay: number analyzed (Participants) | 29
  Week 104: Chromogenic Assay | 51.90 [31.20 to 72.61]
  Week 104: One-Stage Assay: number analyzed (Participants) | 29
  Week 104: One-Stage Assay | 72.91 [47.22 to 98.61]

13. Secondary Outcome: Change From Baseline in Joint Health as Measured by Hemophilia Joint Health Score (HJHS) Instrument at Weeks 24 and 52
Description: A qualified healthcare professional assessed six joints (left ankle, right ankle, left elbow, right elbow, left knee, right knee) scored from 0 to 20 based on: swelling, duration of swelling, muscle atrophy, crepitus on motion, flexion loss, extension loss, joint pain, and strength. Gait was scored (0 to 4) based on walking, stairs, running, hopping on one leg. Total HJHS score = sum of scores from all six joints (left ankle, right ankle, left elbow, right elbow, left knee, right knee) + gait score, ranged from 0 to 124, with the higher score indicated the number equating to more severe joint damage.
Time Frame: Baseline (before infusion on Day 1); Weeks 24 and 52
Population: Dosed analysis population included all participants enrolled in the study and who received the study intervention. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure and "Number Analyzed" signifies number of participants evaluable for at specific timepoints.
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | PF-07055480
Number analyzed (Participants) | 69
Units on a scale
  Change at Week 24 | -1.4 [-2.76 to -0.11]
  Change at Week 52: number analyzed (Participants) | 55
  Change at Week 52 | -2.4 [-3.80 to -0.96]

14. Secondary Outcome: Change From Baseline in Haemophilia Quality of Life Questionnaire (Haem-A-QoL) for Adults Physical Health Domain Score at Weeks 12, 24 and 52
Description: Haem-A-QoL assessed health-related quality of life in adult participants with hemophilia. It contains 46 items with 10 domains that assesses health in the following areas: physical health; feelings; view of self; sports and leisure; work and school; dealing with Haemophilia; treatment; future; family planning; and partnership and sexuality. All items are based on 5-point Likert type scale (1= never, 2= rarely, 3= sometimes, 4= often, 5= all the time). Scoring is performed by averaging non-missing item responses for each domain, then rescaled to be on 0 to 100, with lower scores representing higher quality of life. Total score= was averaged across the 46 items values and then rescaled on 0 to 100, with lower scores representing better quality of life and physical health status. Change from baseline in physical Health domain score was reported in this outcome measure.
Time Frame: Baseline (before infusion on Day 1); Weeks 12, 24 and 52
Population: Dosed analysis population included all participants enrolled in the study and who received the study intervention. All participants reported under "Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row. Here, "Number Analyzed" signifies number of participants evaluable for specified timepoints.
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | PF-07055480
Number analyzed (Participants) | 75
Units on a scale
  Change at Week 12: number analyzed (Participants) | 73
  Change at Week 12 | -13.56 [-18.52 to -8.60]
  Change at Week 24: number analyzed (Participants) | 72
  Change at Week 24 | -14.10 [-19.60 to -8.60]
  Change at Week 52: number analyzed (Participants) | 54
  Change at Week 52 | -9.63 [-15.38 to -3.88]

15. Secondary Outcome: Change From Baseline in Hemophilia Activities List (HAL) Complex Lower Extremity Activities Component Score at Weeks 12, 24 and 52
Description: The HAL was a multiple domain measure of the impact of hemophilia on functional abilities in adults. The 7 domains of this instrument contained 42 items in total, as follows:lying/sitting/kneeling/standing; lower (leg) functioning; upper (arm) functioning; transportation; self-care; household tasks; and sports/leisure. Items were rated on 6-point scale 1 (impossible) to 6 (never) that described difficulty due to hemophilia. HAL total score was calculated according to the Van Genderen scoring algorithm, had a transformed score range from 0 to 100; higher scores indicate better quality of life, that is, less functional limitations in performing tasks. Change from baseline in complex lower extremity activities component score was reported in this outcome measure.
Time Frame: Baseline (before infusion on Day 1); Weeks 12, 24 and 52
Population: Dosed analysis population included all participants enrolled in the study and who receive the study intervention. All participants reported under "Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row. Here, "Number Analyzed" signifies number of participants evaluable for specific timepoints.
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | PF-07055480
Number analyzed (Participants) | 75
Units on a scale
  Change at Week 12: number analyzed (Participants) | 73
  Change at Week 12 | 3.1 [-1.5 to 7.6]
  Change at Week 24: number analyzed (Participants) | 72
  Change at Week 24 | 3.0 [-1.5 to 7.5]
  Change at Week 52: number analyzed (Participants) | 54
  Change at Week 52 | 2.5 [-2.9 to 8.0]

16. Secondary Outcome: ABR for Total Bleeds (Treated and Untreated) Yearly
Description: Treated ABR: An event necessitating administration of coagulation factor within 72 hours of signs or symptoms of bleeding (protocol definition, unless specifically referring to untreated bleed). Untreated ABR: A bleeding event not necessitating administration of coagulation factor within 72 hours of signs and symptoms of bleeding.
Time Frame: Maximum up to 5 years post PF-07055480 infusion
Reporting Status: Not Posted, anticipated posting 2028-10

17. Secondary Outcome: FVIII Activity Levels Yearly
Description: FVIII activity levels will be assessed using one stage assay and chromogenic assay in the central lab.
Time Frame: Maximum up to 5 years post PF-07055480 infusion
Reporting Status: Not Posted, anticipated posting 2028-10

18. Secondary Outcome: AIR of Exogenous FVIII Yearly
Description: AIR: [(Number of exogenous FVIII product infusions for any purpose during the given time period)* 365.25]/ (Number of days of follow-up in the given time period).
Time Frame: Maximum up to 5 years post PF-07055480 infusion
Reporting Status: Not Posted, anticipated posting 2028-10

19. Secondary Outcome: Annualized FVIII Consumption Yearly
Description: Annualized FVIII consumption will be reported in IU/kg and total units (in IU).
Time Frame: Maximum up to 5 years post PF-07055480 infusion
Reporting Status: Not Posted, anticipated posting 2028-10

20. Secondary Outcome: Total (Treated and Untreated) ABR Based on Cause Yearly
Description: Bleeds based on cause were spontaneous (bleeding for no apparent/known reason particularly into the joint, muscles and soft tissue) and traumatic (bleeding event occurring for an apparent/known reason). Bleeds related to a procedure/surgery such as hematomas/bruising which resulted from any surgeries or invasive procedures, or invasive diagnostic were not counted as bleeds. Treated: necessitated administration of coagulation factor within 72 hours of signs or symptoms of bleeding. Untreated: did not necessitate administration of coagulation factor within 72 hours of signs and symptoms of bleeding.
Time Frame: Maximum up to 5 years post PF-07055480 infusion
Reporting Status: Not Posted, anticipated posting 2028-10

21. Secondary Outcome: Treated ABR Based on Cause Yearly
Description: Bleeds based on cause were spontaneous (bleeding for no apparent/known reason particularly into the joint, muscles and soft tissue) and traumatic (bleeding event occurring for an apparent/known reason). Bleeds related to a procedure/surgery such as hematomas/bruising which resulted from any surgeries or invasive procedures, or invasive diagnostic were not counted as bleeds. Treated bleed: necessitated administration of coagulation factor within 72 hours of signs or symptoms of bleeding.
Time Frame: Maximum up to 5 years post PF-07055480 infusion
Reporting Status: Not Posted, anticipated posting 2028-10

22. Secondary Outcome: Total (Treated and Untreated) ABR Based on Location Yearly
Description: Target joint: major joint (hip, elbow, wrist, shoulder, knee, and ankle) with repeated bleeds (3 or more spontaneous bleed into a single joint within 6 month). Joint bleed: bleeding episode by rapid loss of range of motion compared with baseline, associated with pain or an unusual sensation in the joint, swelling. Muscle bleed: bleeding episode into a muscle, determined by imaging study, associated with pain and/or swelling and functional impairment. Treated bleed: necessitated administration of coagulation factor within 72 hrs of sign or symptom of bleeding. Untreated bleed: did not necessitate administration of coagulation factor within 72 hrs of sign and symptom of bleeding.
Time Frame: Maximum up to 5 years post PF-07055480 infusion
Reporting Status: Not Posted, anticipated posting 2028-10

23. Secondary Outcome: Treated ABR Based on Location Yearly
Description: Target joint: major joint (hip, elbow, wrist, shoulder, knee, and ankle) with repeated bleeds (3 or more spontaneous bleed into a single joint within 6 month). Joint bleed: bleeding episode by rapid loss of range of motion compared with baseline, associated with pain or an unusual sensation in the joint, swelling. Muscle bleed: bleeding episode into a muscle, determined by imaging study, associated with pain and/or swelling and functional impairment. Treated bleed: necessitated administration of coagulation factor within 72 hrs of sign or symptom of bleeding.
Time Frame: Maximum up to 5 years post PF-07055480 infusion
Reporting Status: Not Posted, anticipated posting 2028-10

24. Secondary Outcome: Total (Treated and Untreated) ABR Yearly
Description: Bleeds for evaluation included both treated and untreated bleeds. Treated bleed: necessitated administration of coagulation factor within 72 hours of signs or symptoms of bleeding. Untreated bleed: did not necessitate administration of coagulation factor within 72 hours of signs and symptoms of bleeding.
Time Frame: Maximum up to 5 years post PF-07055480 infusion
Reporting Status: Not Posted

25. Secondary Outcome: Treated ABR by Yearly
Description: Treated bleed: bleeding event necessitated administration of coagulation factor within 72 hours of signs or symptoms of bleeding.
Time Frame: Maximum up to 5 years post PF-07055480 infusion
Reporting Status: Not Posted, anticipated posting 2028-10

26. Secondary Outcome: Percentage of Participants Without Bleeds Yearly
Description: as for outcome 24
Time Frame: Maximum up to 5 years post PF-07055480 infusion
Reporting Status: Not Posted, anticipated posting 2028-10

27. Secondary Outcome: Change From Baseline in Joint HJHS Instrument Yearly
Description: A qualified healthcare professional assessed six joints (left ankle, right ankle, left elbow, right elbow, left knee, right knee) scored from 0 to 20 based on: swelling, duration of swelling, muscle atrophy, crepitus on motion, flexion loss, extension loss, joint pain, and strength. Gait was scored (0 to 4) based on walking, stairs, running, hopping on one leg. Total score = sum of scores from all joints + gait score, ranged from 0 to 124, with the higher score indicated the number equating to more severe joint damage.
Time Frame: Baseline (before infusion on Day 1); maximum up to 5 years post PF-07055480 infusion
Reporting Status: Not Posted, anticipated posting 2028-10

28. Secondary Outcome: Change From Baseline in Haem-A-QoL for Adults Physical Health Domain Score Yearly
Description: Haem-A-QoL assessed health-related quality of life in adult participants with hemophilia. It contains 46 items with 10 domains that assesses health in the following areas: physical health; feelings; view of self; sports and leisure; work and school; dealing with Haemophilia; treatment; future; family planning; and partnership and sexuality. All items are based on 5-point Likert type scale (1= never, 2= rarely, 3= sometimes, 4= often, 5= all the time). Scoring is performed by averaging non-missing item responses for each domain, then rescaled to be on 0 to 100, with lower scores representing higher quality of life. Total score= was averaged across the 46 items values and then rescaled on 0 to 100, with lower scores representing better quality of life and physical health status. Change from baseline in physical Health domain score will be reported in this outcome measure.
Time Frame: Baseline (before infusion on Day 1); maximum up to 5 years post PF-07055480 infusion
Reporting Status: Not Posted, anticipated posting 2028-10

29. Secondary Outcome: Change From Baseline in HAL Complex Lower Extremity Activities Component Score Yearly
Description: The HAL was a multiple domain measure of the impact of hemophilia on functional abilities in adults. The 7 domains of this instrument contained 42 items in total, as follows:lying/sitting/kneeling/standing; lower (leg) functioning; upper (arm) functioning; transportation; self-care; household tasks; and sports/leisure. Items were rated on 6-point scale 1 (impossible) to 6 (never) that described difficulty due to hemophilia. HAL total score was calculated according to the Van Genderen scoring algorithm, had a transformed score range from 0 to 100; higher scores indicate better quality of life, that is, less functional limitations in performing tasks. Change from baseline in complex lower extremity activities component score will be reported in this outcome measure.
Time Frame: Baseline (before infusion on Day 1); maximum up to 5 years post PF-07055480 infusion
Reporting Status: Not Posted, anticipated posting 2028-10

30. Secondary Outcome: Treated ABR by Cumulative Follow-up Interval
Description: Treated ABR: an event necessitating administration of coagulation factor within 72 hours of signs or symptoms of bleeding.
Time Frame: Maximum up to 5 years post PF-07055480 infusion
Reporting Status: Not Posted, anticipated posting 2028-10

31. Secondary Outcome: Treated ABR Based on Cause by Cumulative Follow-up Interval
Description: as for outcome 21
Time Frame: Maximum up to 5 years post PF-07055480 infusion
Reporting Status: Not Posted

32. Secondary Outcome: Treated ABR Based on Location by Cumulative Follow-up Interval
Description: Target joint based on location: major joint (hip, elbow, wrist, shoulder, knee, and ankle) with repeated bleeds (3 or more spontaneous bleeds into a single joint within a consecutive 6-month period). Joint bleed: bleeding episode characterized by rapid loss of range of motion as compared with baseline, associated with pain or an unusual sensation in the joint, palpable swelling, and warmth of the skin over the joint. Muscle bleed: bleeding episode into a muscle, determined clinically and/or by imaging study, associated with pain and/or swelling and functional impairment. Treated bleed: necessitated administration of coagulation factor within 72 hrs of sign or symptom of bleeding.
Time Frame: Maximum up to 5 years post PF-07055480 infusion
Reporting Status: Not Posted, anticipated posting 2028-10

33. Secondary Outcome: AIR of Exogenous FVIII by Cumulative Follow-up Interval
Description: as for outcome 18
Time Frame: Maximum up to 5 years post PF-07055480 infusion
Reporting Status: Not Posted, anticipated posting 2028-10

34. Secondary Outcome: Annualized FVIII Consumption by Cumulative Follow-up Interval
Description: Annualized FVIII consumption will be reported in IU/kg and total units (in IU).
Time Frame: Maximum up to 5 years post PF-07055480 infusion
Reporting Status: Not Posted, anticipated posting 2028-10

35. Secondary Outcome: Total (Treated and Untreated) ABR Based on Cause by Cumulative Follow-up Interval
Description: Bleeds based on cause were spontaneous (bleeding for no apparent/known reason particularly into the joint, muscles and soft tissue) and traumatic (bleeding event occurring for an apparent/known reason). Bleeds related to a procedure/surgery such as hematomas/bruising which resulted from any surgeries or invasive procedures, or invasive diagnostic were not counted as bleeds. Treated bleeds: necessitated administration of coagulation factor within 72 hours of signs or symptoms of bleeding. Untreated bleeds: did not necessitate administration of coagulation factor within 72 hours of signs and symptoms of bleeding.
Time Frame: Maximum up to 5 years post PF-07055480 infusion
Reporting Status: Not Posted, anticipated posting 2028-10

36. Secondary Outcome: Total (Treated and Untreated) ABR Based on Location by Cumulative Follow-up Interval
Description: Target joint: major joint (hip, elbow, wrist, shoulder, knee, and ankle) into which repeated bleeds occurred (3 or more spontaneous bleeds into a single joint within a consecutive 6month period). Target joint was considered resolved when there were =<2 bleed into the joint within a 12-month period. Joint bleed: A bleeding episode characterized by rapid loss of range of motion as compared with baseline that was associated with any combination of the following: pain or an unusual sensation in the joint, palpable swelling, and warmth of the skin over the joint. Muscle bleed: an episode of bleeding into a muscle, determined clinically and/or by imaging studies, generally associated with pain and/or swelling and functional impairment. Treated bleed: necessitated administration of coagulation factor within 72 hrs of sign or symptom of bleeding. Untreated bleed: did not necessitate administration of coagulation factor within 72 hrs of sign and symptom of bleeding.
Time Frame: Maximum up to 5 years post PF-07055480 infusion
Reporting Status: Not Posted, anticipated posting 2028-10

37. Secondary Outcome: Percentage of Participants Without Bleeds by Cumulative Follow-up Interval
Description: as for outcome 24
Time Frame: Maximum up to 5 years post PF-07055480 infusion
Reporting Status: Not Posted, anticipated posting 2028-10

38. Secondary Outcome: Total ABR (Treated and Untreated) by Cumulative Follow-up Interval
Description: Bleeds for evaluation included both treated and untreated bleeds. Treated bleed: bleeding event necessitated administration of coagulation factor within 72 hours of signs or symptoms of bleeding. Untreated bleed: bleeding event did not necessitate administration of coagulation factor within 72 hours of signs and symptoms of bleeding.
Time Frame: Maximum up to 5 years post PF-07055480 infusion
Reporting Status: Not Posted, anticipated posting 2028-10

39. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Severe AEs
Description: An AEs was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Severe AEs: An event that prevented normal everyday activities. Severe was a category utilized for rating the intensity of an event, and both AEs and serious adverse events (SAEs) could be assessed as severe.
Time Frame: From Day 1 up to 104 weeks after last dose of PF-07055480 (maximum for 44.4 months)
Population: Safety population included all participants enrolled in the study who received the study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07055480
Number analyzed (Participants) | 75
Participants
  AEs | 74
  Severe AEs | 7

40. Secondary Outcome: Number of Participants With AEs of Special Interest
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. AESI included all medically important events that were reported as a serious adverse events (SAE), and any clinical reported thrombotic event or hypersensitivity/infusion-related reactions events assessed as non-serious AEs.
Time Frame: From Day 1 up to 104 weeks after last dose of PF-07055480 (maximum for 44.4 months)
Population: Safety population included all participants enrolled in the study who received the study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07055480
Number analyzed (Participants) | 75
Participants | 70

41. Secondary Outcome: Number of Participants With Positive Antibodies Against Adeno-Associated Virus Vector 6 (AAV6) Capsid Protein
Description: Number of participants with positive antibodies against AAV6 Capsid protein will be reported in this outcome measure.
Time Frame: Maximum up to 5 years post PF-07055480 infusion
Reporting Status: Not Posted, anticipated posting 2028-10

42. Secondary Outcome: Number of Participants With T-cell Responses Against AAV6 Capsid and FVIII by Elispot Assay
Description: The enzyme linked immune spot (ELISPOT) assay is a highly sensitive quantitative immunoassay for measuring relevant parameters of T cell activation (the frequency of cytokine-secreting cells at the single-cell level) on peripheral blood mononuclear cells (PBMC). T cell responses to AAV6 and FVIII will be evaluated at baseline and during study follow up, if corticosteroid treatment is needed for a suspected T-cell response.
Time Frame: Maximum up to 5 years post PF-07055480 infusion
Reporting Status: Not Posted, anticipated posting 2028-10

43. Secondary Outcome: Number of Participants With FVIII Inhibitors Status by Bethesda Assessment
Description: Nijmegen Bethesda assay will be used to assess the presence of FVIII inhibitors (Inhibitory antibodies against FVIII that neutralize the clotting activity of FVIII). Positive refers to FVIII inhibitor levels by inhibitor assay results >=0.6 Bethesda units per milliliter (BU/mL).
Time Frame: Maximum up to 5 years post PF-07055480 infusion
Reporting Status: Not Posted, anticipated posting 2028-10

ADVERSE EVENTS:
Time Frame: From Day 1 up to 104 weeks after last dose of PF-07055480 (maximum for 44.4 months)
Description: Same event may appear as both non-SAE and a serious AE. However, what is presented are distinct events. An event may be categorized as SAE in one participant and as non-SAE in another participant, or one participant may have experienced both. SAS included all participants enrolled in the study and who received the study intervention.
Arm/Group | PF-07055480
All-Cause Mortality (participants affected / at risk) | 0/75
Serious Adverse Events (participants affected / at risk) | 15/75
Other Adverse Events (participants affected / at risk) | 70/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-07055480 (N=75)
Ocular hyperaemia (Eye disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Chills (General disorders) | 1
Facial pain (General disorders) | 1
Pyrexia (General disorders) | 5
Swelling face (General disorders) | 1
Immune-mediated adverse reaction (Immune system disorders) | 1
COVID-19 (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Myelitis (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Muscle rupture (Injury, poisoning and procedural complications) | 1
Anti factor VIII antibody positive (Investigations) | 2
Transaminases increased (Investigations) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 1
Ductal adenocarcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-07055480 (N=75)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 4
Tachycardia (Cardiac disorders) | 6
Abdominal pain upper (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 10
Dyspepsia (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 23
Vomiting (Gastrointestinal disorders) | 8
Asthenia (General disorders) | 5
Chills (General disorders) | 16
Fatigue (General disorders) | 11
Pain (General disorders) | 4
Pyrexia (General disorders) | 45
COVID-19 (Infections and infestations) | 9
Influenza (Infections and infestations) | 8
Nasopharyngitis (Infections and infestations) | 6
Upper respiratory tract infection (Infections and infestations) | 11
Alanine aminotransferase increased (Investigations) | 37
Aspartate aminotransferase increased (Investigations) | 13
Coagulation factor VIII level decreased (Investigations) | 8
Coagulation factor VIII level increased (Investigations) | 7
Factor VIII activity decreased (Investigations) | 7
Factor VIII activity increased (Investigations) | 18
Transaminases increased (Investigations) | 4
Iron deficiency (Metabolism and nutrition disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 16
Back pain (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Dizziness (Nervous system disorders) | 6
Headache (Nervous system disorders) | 38
Hypoaesthesia (Nervous system disorders) | 4
Insomnia (Psychiatric disorders) | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5
Acne (Skin and subcutaneous tissue disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 4
Hypertension (Vascular disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-11-15): https://cdn.clinicaltrials.gov/large-docs/54/NCT04370054/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-09): https://cdn.clinicaltrials.gov/large-docs/54/NCT04370054/SAP_001.pdf